CLINICAL TRIAL: NCT00659295
Title: A Multicentre, Open Label, Nonrandomised, Non-interventional, Observational, Safety Study in Subjects Using Insulin Detemir for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus: The PREDICTIVE™ Study: Predictable Results and Experience in Diabetes Through Intensification and Control to Target: an International Variability Evaluation
Brief Title: Observational Study to Evaluate the Safety of Levemir® in Diabetes
Acronym: PREDICTIVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1677
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Prescription of insulin detemir (Levemir®) according to local approved labelling by prescribing physician in a normal clinical practice to patients with type 1 diabetes, including newly diagnosed patients who have never received insulin or analogue treatment.
  Interventions: Drug: insulin detemir
- Type 2 diabetes: Prescription of insulin detemir (Levemir®) according to local approved labelling by prescribing physician in a normal clinical practice to patients with type 1 diabetes, including newly diagnosed patients who have never received insulin or analogue treatment.
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of a normal clinical practice.

SUMMARY:
This study is conducted in Africa, Asia, Europe, Japan and South America. The aim of this observational study is to evaluate the incidence of serious adverse reactions (SARs) while using Levemir® (insulin detemir) under normal clinical practice conditions.

Study conducted globally in 26 countries. Some countries participated in the study for only 3 months (Austria, Brazil, Denmark, Germany, Israel, Lebanon, Slovenia, Russia, and Turkey), while others extended their participation to 6 (Belgium/Luxembourg, Czech Republic, Greece, India, Italy, Netherlands, Saudi Arabia, South Africa, South Korea, Sweden, Tunisia, and United Kingdom/Ireland) and 12 months (Finland, France, and Japan), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age according to approved label in each country and physician discretion
* Type 1 or 2 diabetes
* Recently started treatment with insulin detemir at the discretion of the investigator. Before initiation of insulin detemir they should not have been treated with insulin
* Selection at the discretion of the physician

Exclusion Criteria:

* Current treatment with Levemir® (insulin detemir)
* Previously enrolled in the study
* Hypersensitivity to Levemir® (insulin detemir)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from both general and speciality practice settings who have been deemed appropriate to receive Levemir® (insulin detemir) as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 51170 (Actual)
Dates: Start 2004-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (13):
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Copenhagen S, Denmark
- Novo Nordisk Investigational Site, Espoo, Finland
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Vouliagment, Greece
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Malmo, Sweden
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Dornhorst A, Luddeke HJ, Honka M, Ackermann RW, Merilainen M, Gallwitz B, Sreenan S; PREDICTIVE Study Group. Safety and efficacy of insulin detemir basal-bolus therapy in type 1 diabetes patients: 14-week data from the European cohort of the PREDICTIVE study. Curr Med Res Opin. 2008 Feb;24(2):369-76. doi: 10.1185/030079908x260835. PMID 18096110
- [Result] Honka M. [Results of the PREDICTIVE project in the Czech Republic]. Vnitr Lek. 2008 Apr;54(4):361-7. Czech. PMID 18630615
- [Result] Dornhorst A, Luddeke HJ, Koenen C, Merilainen M, King A, Robinson A, Sreenan S; PREDICTIVE Study Group. Transferring to insulin detemir from NPH insulin or insulin glargine in type 2 diabetes patients on basal-only therapy with oral antidiabetic drugs improves glycaemic control and reduces weight gain and risk of hypoglycaemia: 14-week follow-up data from PREDICTIVE. Diabetes Obes Metab. 2008 Jan;10(1):75-81. doi: 10.1111/j.1463-1326.2007.00816.x. Epub 2007 Nov 22. PMID 18034846
- [Result] Dornhorst A, Luddeke HJ, Sreenan S, Koenen C, Hansen JB, Tsur A, Landstedt-Hallin L. Safety and efficacy of insulin detemir in clinical practice: 14-week follow-up data from type 1 and type 2 diabetes patients in the PREDICTIVE European cohort. Int J Clin Pract. 2007 Mar;61(3):523-8. doi: 10.1111/j.1742-1241.2007.01316.x. PMID 17313628
- [Result] Dornhorst A, Luddeke HJ, Sreenan S, Kozlovski P, Hansen JB, Looij BJ, Meneghini L; PREDICTIVE Study Group. Insulin detemir improves glycaemic control without weight gain in insulin-naive patients with type 2 diabetes: subgroup analysis from the PREDICTIVE study. Int J Clin Pract. 2008 Apr;62(4):659-65. doi: 10.1111/j.1742-1241.2008.01715.x. PMID 18324957
- [Result] Luddeke HJ, Sreenan S, Aczel S, Maxeiner S, Yenigun M, Kozlovski P, Gydesen H, Dornhorst A; PREDICTIVE Study Group. PREDICTIVE- a global, prospective observational study to evaluate insulin detemir treatment in types 1 and 2 diabetes: baseline characteristics and predictors of hypoglycaemia from the European cohort. Diabetes Obes Metab. 2007 May;9(3):428-34. doi: 10.1111/j.1463-1326.2006.00677.x. PMID 17391171
- [Result] Sreenan S, Virkamaki A, Zhang K, Hansen JB; PREDICTIVE study group. Switching from NPH insulin to once-daily insulin detemir in basal-bolus-treated patients with diabetes mellitus: data from the European cohort of the PREDICTIVE study. Int J Clin Pract. 2008 Dec;62(12):1971-80. doi: 10.1111/j.1742-1241.2008.01939.x. PMID 19166444
- [Result] Palmer JL, Goodall G, Nielsen S, Kotchie RW, Valentine WJ, Palmer AJ, Roze S. Cost-effectiveness of insulin aspart versus human soluble insulin in type 2 diabetes in four European countries: subgroup analyses from the PREDICTIVE study. Curr Med Res Opin. 2008 May;24(5):1417-28. doi: 10.1185/030079908x297295. Epub 2008 Apr 8. PMID 18400145
- [Result] Valentine WJ, Goodall G, Aagren M, Nielsen S, Palmer AJ, Erny-Albrecht K. Evaluating the cost-effectiveness of therapy conversion to insulin detemir in patients with type 2 diabetes in Germany: a modelling study of long-term clinical and cost outcomes. Adv Ther. 2008 Jun;25(6):567-84. doi: 10.1007/s12325-008-0069-z. PMID 18568451
- [Result] Hermansen K, Lund P, Clemmensen K, Breum L, Kleis Moller M, Mette Rosenfalck A, Christiansen E; Danish PREDICTIVE study group. 3-Month Results from Denmark within the Globally Prospective and Observational Study to Evaluate Insulin Detemir Treatment in Type 1 and Type 2 Diabetes: The PREDICTIVE Study. Rev Diabet Stud. 2007 Summer;4(2):89-97. doi: 10.1900/RDS.2007.4.89. Epub 2007 Aug 10. PMID 17823693
- [Result] Fontaine P, Gin H, Pinget M, Thivolet C, Hanaire H, Robert JJ, Marre M, Venkatanarasimhachar S. Effect of insulin detemir dose frequency on clinical outcomes in patients with diabetes in PREDICTIVE. Adv Ther. 2009 May;26(5):535-51. doi: 10.1007/s12325-009-0033-6. Epub 2009 Jun 2. PMID 19513632
- [Result] Hermansen K, Dornhorst A, Sreenan S. Observational, open-label study of type 1 and type 2 diabetes patients switching from human insulin to insulin analogue basal-bolus regimens: insights from the PREDICTIVE study. Curr Med Res Opin. 2009 Nov;25(11):2601-8. doi: 10.1185/03007990903262885. PMID 19739940
- [Result] Niskanen L, Virkamaki A, Hansen JB, Saukkonen T. Fasting plasma glucose variability as a marker of nocturnal hypoglycemia in diabetes: evidence from the PREDICTIVE study. Diabetes Res Clin Pract. 2009 Nov;86(2):e15-8. doi: 10.1016/j.diabres.2009.08.005. Epub 2009 Sep 10. PMID 19747748
- [Result] Yenigun M, Honka M. Switching patients from insulin glargine-based basal-bolus regimens to a once daily insulin detemir-based basal-bolus regimen: results from a subgroup of the PREDICTIVE study. Int J Clin Pract. 2009 Mar;63(3):425-32. doi: 10.1111/j.1742-1241.2008.01973.x. PMID 19222627
- [Result] Perriello G, Caputo S, De Pergola G, Di Carlo A, Grassi G, Lapolla A, Pata P, Solerte SB, Zaccardi F. Improved glycemic control with weight loss and a low risk of hypoglycemia with insulin detemir: insights from the Italian cohort of the PREDICTIVE study after 6-month observation in type 2 diabetic subjects. Expert Opin Pharmacother. 2011 Nov;12(16):2449-55. doi: 10.1517/14656566.2011.626766. PMID 21988213
- [Result] Yang L, Christensen T, Sun F, Chang J. Cost-effectiveness of switching patients with type 2 diabetes from insulin glargine to insulin detemir in Chinese setting: a health economic model based on the PREDICTIVE study. Value Health. 2012 Jan-Feb;15(1 Suppl):S56-9. doi: 10.1016/j.jval.2011.11.018. PMID 22265068
- [Result] Sreenan S, Andersen M, Thorsted BL, Wolden ML, Evans M. Increased Risk of Severe Hypoglycemic Events with Increasing Frequency of Non-severe Hypoglycemic Events in Patients with Type 1 and Type 2 Diabetes. Diabetes Ther. 2014 Dec;5(2):447-58. doi: 10.1007/s13300-014-0075-x. Epub 2014 Jul 15. PMID 25023521
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted globally in 26 countries. Some countries participated for only 3 months, while others extended their participation to 6 and 12 months, respectively.
Pre-assignment Details: Subjects with type 1 or type 2 diabetes including newly diagnosed subjects who had never received insulin or an insulin analogue at the prescribing physician's discretion.
Period: Overall Study
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Started | 13529 | 37641
Completed | 10821 | 32038
Not Completed | 2708 | 5603

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 1 Diabetes | Type 2 Diabetes | Total
Number analyzed (Participants) | 13529 | 37641 | 51170
Age, Continuous [Mean (Standard Deviation); unit: years] — Age: 3 months' participation
  years
    Austria, n=331, 430 | 41.9 (13.8) | 60.8 (11.5) | 52.6 (12.5)
    Brazil, n=962, 1136 | 29.6 (15.5) | 60.3 (12.9) | 46.2 (14.1)
    Denmark, n=312, 77 | 45.6 (13.3) | 61.4 (10.9) | 48.7 (12.8)
    Germany, n=2640, 7526 | 45.0 (15.7) | 62.3 (10.4) | 57.8 (11.8)
    Israel, n=295, 722 | 36.5 (20.0) | 60.2 (11.1) | 53.3 (13.7)
    Lebanon, n=63, 192 | 27.6 (10.3) | 58.2 (11.6) | 50.6 (11.3)
    Russia, n=1121, 2515 | 28.5 (15.8) | 58.7 (9.8) | 49.4 (11.6)
    Slovenia, n=91, 209 | 42.3 (14.5) | 59.1 (10.0) | 54.0 (11.4)
    Turkey, n=622, 2132 | 28.9 (15.2) | 55.9 (10.5) | 49.8 (11.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age: 6 months' participation
  years
    Belgium/Luxembourg, n=330, 38 | 45.2 (15.4) | 62.4 (9.6) | 47.0 (14.8)
    Czech Republic, n=861, 820 | 45.3 (16.8) | 59.4 (10.7) | 52.2 (13.8)
    Greece, n=125, 923 | 31.6 (16.3) | 64.9 (11.2) | 60.9 (11.8)
    India, n=142, 3162 | 31.4 (17.0) | 52.6 (10.1) | 51.7 (10.4)
    Italy, n=177, 1297 | 44.6 (16.0) | 64.9 (9.8) | 62.5 (11.5)
    Netherlands, n=92, 324 | 39.9 (16.6) | 59.7 (13.0) | 55.3 (13.8)
    Saudi Arabia, n=104, 503 | 25.0 (13.1) | 50.0 (10.5) | 45.7 (10.9)
    South Africa, n=207, 247 | 33.6 (16.0) | 53.3 (11.9) | 44.3 (13.8)
    South Korea, n=224, 8854 | 36.0 (16.0) | 56.9 (12.4) | 56.4 (12.5)
    Sweden, n=553, 95 | 42.0 (17.5) | 61.3 (11.2) | 44.8 (16.6)
    Tunisia, n=21, 316 | 24.5 (15.9) | 57.6 (11.1) | 55.5 (11.4)
    United Kingdom/Ireland, n=2292, 1832 | 35.5 (17.6) | 59.2 (11.7) | 46.0 (15.0)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age: 12 months' participation
  years
    Finland, n=809, 249 | 41.9 (14.3) | 58.8 (10.7) | 45.9 (13.5)
    France, n=641, 1127 | 47.1 (16.1) | 62.6 (11.9) | 57.0 (13.4)
    Japan, n=490, 2801 | 50.5 (16.1) | 61.9 (12.8) | 60.2 (13.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 6865 | 19175 | 26040
  Male | 6658 | 18453 | 25111
  Not specified | 6 | 13 | 19
Duration of diabetes (3 months' participation) [Mean (Standard Deviation); unit: years]
  Austria, n=330, 428 | 18.5 (13.6) | 12.5 (8.5) | 15.1 (10.7)
  Brazil, n=959, 1141 | 12.6 (9.7) | 13.7 (9.0) | 13.2 (9.3)
  Denmark, n=312, 76 | 20.4 (12.6) | 11.8 (6.6) | 18.7 (11.4)
  Germany, n=2607, 7468 | 17.2 (12.5) | 10.6 (7.2) | 12.3 (8.6)
  Israel, n=286, 721 | 14.3 (12.4) | 15.7 (9.1) | 15.3 (10.0)
  Lebanon, n=63, 192 | 11.4 (7.7) | 12.2 (7.1) | 12.0 (7.2)
  Russia, n=1112, 2509 | 8.5 (8.2) | 9.5 (5.8) | 9.2 (6.5)
  Slovenia, n=90, 208 | 18.1 (13.0) | 13.7 (8.0) | 15.0 (9.5)
  Turkey, n=612, 2127 | 8.2 (6.7) | 10.6 (6.6) | 10.1 (6.6)
Duration of diabetes (6 months' participation) [Mean (Standard Deviation); unit: years]
  Belgium/Luxembourg, n=329, 38 | 17.7 (12.3) | 14.0 (9.2) | 17.3 (12.0)
  Czech Republic, n=856, 807 | 14.5 (11.1) | 12.8 (7.8) | 13.7 (9.5)
  Greece, n=129, 956 | 11.9 (9.9) | 13.4 (7.6) | 13.2 (7.9)
  India, n=139, 3178 | 6.6 (6.2) | 8.5 (5.5) | 8.4 (5.5)
  Italy, n=175, 1292 | 14.6 (11.6) | 14.7 (8.6) | 14.7 (9.0)
  Netherlands, n=88, 318 | 16.0 (14.5) | 9.6 (6.9) | 11.0 (8.5)
  Saudi Arabia, n=96, 494 | 7.2 (6.3) | 9.1 (5.6) | 8.8 (5.7)
  South Africa, n=196, 243 | 11.3 (9.4) | 9.9 (7.4) | 10.5 (8.3)
  South Korea, n=214, 8701 | 9.4 (7.7) | 10.1 (6.8) | 10.1 (6.8)
  Sweden, n=547, 96 | 19.6 (14.2) | 13.6 (7.4) | 18.7 (13.2)
  Tunisia, n=21, 316 | 8.2 (7.7) | 11.5 (6.4) | 11.3 (6.5)
  United Kingdom/Ireland, n=2260, 1827 | 15.2 (12.3) | 11.3 (7.7) | 13.5 (10.2)
Duration of diabetes (12 months' participation) [Mean (Standard Deviation); unit: years]
  Finland, n=796, 245 | 19.8 (12.3) | 13.3 (7.6) | 18.3 (11.2)
  France, n=628, 1117 | 17 (12) | 14.6 (8.9) | 15.5 (10)
  Japan, n=420, 2240 | 12.1 (10) | 14.2 (8.9) | 13.9 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Reactions, Including Major Hypoglycaemic Events
Description: The incidence of serious adverse reactions (SARs), including major hypoglycaemic events, during 3 months of insulin detemir therapy for all countries participating in the study, and during 6 and 12 months of insulin detemir therapy for some of the participating countries. The three sub-groups were mutually exclusive. Physicians did not report all major hypoglycaemic events as SARs. The values in the SAE table are SARs including only those major hypoglycaemic events that were reported as SARs by physicians.
Time Frame: Months 0-12
Population: FAS (Full Analysis Set) consists of all patients with a baseline visit who were prescribed insulin detemir at least once
Measure: Number; unit: participants
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 13529 | 37641
participants
  3 months sub-group | 186 | 93
  6 months sub-group | 208 | 112
  12 months sub-group | 109 | 48

ADVERSE EVENTS:
Time Frame: Over 3, 6 and 12 months, respectively, depending on the participating country
Description: Full Analysis Set. This is a non-interventional study. According to the primary endpoint/outcome measure, the serious events collected in all countries are Serious Drug Reactions only, and not Serious Adverse Events and other adverse events
Arm/Group | Type 1 Diabetes | Type 2 Diabetes
Serious Adverse Events (participants affected / at risk) | 130/13529 | 80/37641
Other Adverse Events (participants affected / at risk) | 0/13529 | 0/37641
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Diabetes (N=13529) | Type 2 Diabetes (N=37641)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Injection site stinging (General disorders) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blister (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limp injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increase (Investigations) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood glucose decrease (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 (7) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 66 (73) | 33 (34)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 8 (8) | 0 (0)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coma acidotic (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 21 (21) | 7 (11)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 6 (6) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Transmyocardial revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the physician's right to publish the entire results of the trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.